CLINICAL TRIAL: NCT03466320
Title: An Open-label, Phase I/II Study to Assess the Safety and Clinical Activity of NKR-2 Treatment Administration After a Non-myeloablative Preconditioning Chemotherapy in Relapse/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome Patients.
Brief Title: DEPLETHINK - LymphoDEPLEtion and THerapeutic Immunotherapy With NKR-2
Acronym: DEPLETHINK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-N2T-005
Record Dates: First submitted 2018-02-16; First posted 2018-03-15 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: AML; MDS
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase I Dose Escalation Segment 1 - T7-DL1 (Experimental): Preconditioning (consisting in cyclophosphamide 300 mg/m² and fludarabine 30 mg/m² daily {CYFLU}) at days -9, -8 and -7.
  Dose 1: 1x108 NKR-2 (adjusted at 1.5x106 NKR-2/kg for patients with body weight ≤ 65 kg) administered at 7 days (T7) after the end of the preconditioning regimen
  Interventions: Biological: NKR-2
- Phase I Dose Escalation Segment 1 - T3-DL1 (Experimental): Preconditioning (consisting in cyclophosphamide 300 mg/m² and fludarabine 30 mg/m² daily {CYFLU}) at days -5, -4 and -3.
  Dose 1: 1x108 NKR-2 (adjusted at 1.5x106 NKR-2/kg for patients with body weight ≤ 65 kg) administered at 3 days (T3) after the end of the preconditioning regimen
  Interventions: Biological: NKR-2
- Phase I Dose Escalation Segment 1 - T3-DL2 (Experimental): Preconditioning (consisting in cyclophosphamide 300 mg/m² and fludarabine 30 mg/m² daily {CYFLU}) at days -5, -4 and -3.
  Dose 2: 3x108 NKR-2 (adjusted at 4.6x106 NKR-2/kg for patients with body weight ≤ 65 kg) administered at 3 days (T3) after the end of the preconditioning regimen
  Interventions: Biological: NKR-2
- Phase I Dose Escalation Segment 1 - T3-DL3 (Experimental): Preconditioning (consisting in cyclophosphamide 300 mg/m² and fludarabine 30 mg/m² daily {CYFLU}) at days -5, -4 and -3.
  Dose 3: 1x109 NKR-2 (adjusted at 1.5x107 NKR-2/kg for patients with body weight ≤ 65 kg) administered at 3 days (T3) after the end of the preconditioning regimen
  Interventions: Biological: NKR-2
- Phase I Dose Escalation - extension (Experimental): This extension segment will enroll more patients (to reach 9 evaluable patients in total) to further evaluate the selected treatment regimen, i.e., the recommended NKR-2 dose (1x108 or 3x108 or 1x109NKR-2/injection) with the CYFLU preconditioning treatment administered at the recommended interval (T3 or T7) prior to NKR-2 administration.
  Interventions: Biological: NKR-2
- Phase II Segment 1 (Experimental): This extension segment will enroll more patients (to reach 13 evaluable patients in total) to further evaluate the selected treatment regimen, i.e., the recommended NKR-2 dose (1x108 or 3x108 or 1x109NKR-2/injection) with the CYFLU preconditioning treatment administered at the recommended interval (T3 or T7) prior to NKR-2 administration.
  Interventions: Biological: NKR-2
- Phase II Segment 2 (Experimental): Enrollment in the Phase II part of the study will be divided in 2 consecutive segments, with 13 patients in total in the segment 1 and 30 new patients in segment 2 (43 patients in total) if the study is not terminated due to futility, according a Simon's two-stage optimal design
  Interventions: Biological: NKR-2

INTERVENTIONS:
Biological: NKR-2 — This Phase I study will explore the hypothesis that the administration of modified T-cells targeting NKG2D-ligands expressed by AML/MDS cells, after a prior nonmyeloablative preconditioning treatment, in patients refractory to and/or relapsing after prior therapies, is safe and, considering the poor outcomes and lack of therapeutic strategies for this patient population, may have a strategic advantage over current approaches and provide potential clinical benefit.
  Other Names: cyclophosphamide 300 mg/m²; fludarabine 30 mg/m²

SUMMARY:
This open-label Phase I study aims at assessing primarily the safety of the NKR-2 treatment administered after a non-myeloablative preconditioning regimen in r/r AML/MDS patients.

This Phase I study will contain two different sequential segments. The first segment will determine the recommended investigational treatment option (schedule of preconditioning and NKR-2 dose) and the second segment will expand to a larger number of r/r AML/MDS patients.

DETAILED DESCRIPTION:
This open-label Phase I/II study aims at assessing primarily the safety and the clinical activity of the NKR-2 treatment administered after a non-myeloablative preconditioning regimen in r/r AML/MDS patients.

The Phase I part of the study will contain two different sequential segments. The first segment (dose escalation segment) will determine the recommended investigational treatment option (schedule of preconditioning and NKR-2 dose) and the second segment (extension segment) will expand to a larger number of r/r AML/MDS patients.

The Phase II part of the study will also contain two sequential segments, assessing the clinical activity of the NKR-2 treatment administrated as per the recommended investigational treatment option (schedule of preconditioning and NKR-2 dose).

The Phase I dose escalation segment will evaluate the preconditioning regimen consisting in cyclophosphamide 300 mg/m² and fludarabine 30 mg/m² daily (CYFLU) administrated 3 consecutive days at a specific interval prior to the NKR 2 administration. This segment is divided into four sequential cohorts to evaluate respectively:

* Two different intervals between the preconditioning regimen and the NKR-2 administration i.e. NKR-2 administered 3 days (T3) or 7 days (T7) after the end of the preconditioning regimen,
* Three different NKR-2 dose-levels i.e. dose-level 1 (1x108 NKR 2/injection), dose-level 2 (3x108 NKR-2/injection) and dose-level 3 (1x109 NKR-2/injection).

The Phase I extension segment will enroll more r/r AML/MDS patients (to reach 9 evaluable patients in total) to further evaluate the recommended NKR-2 dose (1x108, 3x108 or 1x109 NKR-2/injection) administered at the recommended interval (T3 or T7) after the CYFLU preconditioning.

The Phase II will enroll more r/r AML/MDS patients (13 patients in total in the segment 1 and 30 new patients in the segment 2) to further evaluate the recommended NKR-2 dose (1x108, 3x108 or 1x109 NKR-2/injection) administered at the recommended interval (T3 or T7) after the CYFLU preconditioning to assess the clinical activity.

Each patient will receive a single administration of NKR-2 following the preconditioning regimen. Depending on the clinical response as evaluated at the first tumor assessment, scheduled three weeks after NKR-2 administration, three situations may arise:

* If the patient is presenting a complete remission, partial remission, or stable disease, and meets all criteria for a consolidation cycle, then three new injections of NKR-2 at the recommended dose defined in the ongoing THINK study (THINK RecD), without prior preconditioning, will be administered with a two weeks interval,
* If the patient is in PD, or does not meet all criteria for the consolidation cycle he/she will not receive any other NKR-2 injection but will follow other visits as scheduled.

For each patient who received at least one NKR-2 administration, the overall study duration will be 15 years after first NKR-2 administration.

The duration of the administration phase and treatment follow-up will be 24 months.

Patients will be asked to complete a total of maximum 20 visits during the treatment administration phase, and maximum 6 visits during the treatment follow-up phase. During the long-term safety follow-up, yearly visits will be scheduled (up to Y15).

Rationale for the study:

NKR-2 has the potential to treat many distinct tumor-types because of a broad expression and important prevalence of the NKG2D ligands expression in various tumor types including in r/r AML/MDS. This Phase I study will explore the hypothesis that the administration of modified T-cells targeting NKG2D-ligands expressed by AML/MDS cells, after a prior nonmyeloablative preconditioning treatment, in patients refractory to and/or relapsing after prior therapies, is safe and, considering the poor outcomes and lack of therapeutic strategies for this patient population, may have a strategic advantage over current approaches and provide potential clinical benefit.

Objectives of the study:

Primary

To document and characterize:

* The safety of the NKR-2 treatment administration in r/r AML/MDS patients after a non-myeloablative preconditioning. (Phase I part)
* The objective response rate (ORR) post the first NKR-2 administration. (Phase II part)

Secondary

To document and characterize:

* The NKR-2 peripheral blood kinetics post-administration,
* Indicators of clinical activity,
* Additional indicators of safety.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have signed the written ICF and must accept that, beyond the treatment period, and the treatment follow-up period, he/she will have to be monitored for a Long-Term Safety Follow-Up (LTSFU) for up to 15 years after enrollment.
2. Both men and women of all races and ethnic groups are eligible.
3. The patient must be ≥ 18 and ≤ 75 years old at the time of signing the ICF.
4. The patient must not be eligible for standard of care therapy and have one of the following hematological malignancy:

4.a. A confirmed relapsed or refractory acute myeloid leukemia (AML) (i.e. ≥ 5% blasts in bone marrow or in peripheral blood) after at least one prior therapy defined as either

* Recurrence of disease after a first complete remission (CR1) and not eligible for a second course of induction therapy, or
* Recurrence of disease after a second complete remission (CR2), or
* Failure to achieve CR after induction chemotherapy. Note: Patient with AML M3 are excluded. 4.b. A confirmed myelodysplastic syndrome (MDS) with:
* Revised International Prognostic Scoring System (R-IPSS) criteria for Intermediate, High-risk or Very High-risk disease or refractory anemia with excess blasts by WHO (i.e. ≥ 5% blasts in bone marrow or ≥ 2% blasts in peripheral blood) or MDS with TP53 mutation as detected by next-generation sequencing (NGS).
* Failure of prior treatment with at least 4 cycles of azacitidine or decitabine defined as no response to treatment, loss of response at any time point, or progressive disease/intolerance to therapy.

  5. The absolute peripheral blast count should be < 15,000/L. 6. The patient must have evaluable disease defined by:
* Revised Recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, for AML patients,
* IWG 2006 Uniform Response Criteria for patients with Higher-Risk MDS. 7. The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status below or equal to 2.

  8. The patient must have adequate hepatic and renal functions as assessed by standard laboratory criteria 9. The patient must have a left ventricular ejection fraction (LVEF) of more than or equal to 40%, as determined by echocardiography or a multigated acquisition (MUGA) scan.

  10. The patient must have a good pulmonary function with a Forced Expiratory Volume in the first second (FEV-1)/Forced Vital Capacity (FVC) more than or equal to 0.7 with FEV-1 more than or equal to 50% predicted (GOLD 1 or 2 severity) as determined by the spirometry performed at baseline , unless related to the AML/MDS disease as judged by the Investigator.

  11. Women of child-bearing potential and men must agree to use effective contraception before, during and for at least 2 months after the last study treatment administration.

  12. The patient must, in the opinion of the Investigator, be able to adhere with the study visit schedule and all study procedures described in this protocol.

Exclusion Criteria:

1. The patient has a confirmed or history of tumor involvement in the central nervous system (CNS).
2. Patients who have received any cancer therapy (investigational agent or not), including but not limited to chemotherapy, small molecules, monoclonal antibodies (e.g., immune checkpoint blockade therapies), or radiotherapy within 2 weeks before the planned day for the apheresis (Day -21)
3. Patients who are planned to receive, concurrently receiving or have received any investigational agent within 3 weeks before the planned day for the first NKR-2 administration (Day 1).
4. Patient is under systemic immunosuppressive drugs, unless specific cases authorized per protocol.
5. Patients who have received prior allogeneic stem cell transplantation or chimeric antigen receptor therapy.
6. Patients who are presenting persistent toxicities greater than or equal to CTCAE grade 2 caused by previous cancer therapy (except for clinically non-significant toxicities, such as alopecia).
7. Presence of any indwelling catheter or drain (e.g., percutaneous nephrostomy tube, indwelling foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter) may be permissible unless they have a catheter-associated infection that cannot be cleared with antibiotics. Ommaya reservoirs and dedicated central venous access catheters such as a Port-a-Cath, peripherally inserted central catheter, or Hickman catheter are permitted.
8. Patients who underwent major surgery within 4 weeks before the planned day for the first NKR-2 administration (Day 1).
9. Patients who have received a live vaccine ≤ 6 weeks prior to each NKR 2 administration.
10. Patients with uncontrolled intercurrent illness or serious uncontrolled medical disorder including, but not limited to evidence of active pneumonitis on screening chest imaging, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia history (or evidenced after the electrocardiogram planned at screening) and/or pronounced disturbances of the electrical conduction system of the heart, or significant thromboembolic events.
11. Patients with significant disorder of coagulation or receiving treatment with warfarin derivatives or heparin.
12. Patients who have active infections including, but not limited to viral, bacterial or fungal infections necessitating use of antibiotics/antivirals/antifungal treatment (prophylaxis is acceptable).
13. Patients who are known to be positive or screened positive for hepatitis B (HBsAg positive) or C (anti-HCV positive).
14. Patients who are known to be positive or screened positive for the human immunodeficiency virus (HIV).
15. Patients with a family history of congenital or hereditary immunodeficiency.
16. Patients with a history of allergic reactions or hypersensitivity attributed to Human serum albumin or Plasma-lyte A.
17. Patient with history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis and/or active or acute exacerbation of chronic obstructive pulmonary disease (COPD).
18. Patients on supplemental home oxygen.
19. Patients with history of any autoimmune disease including, but not limited to inflammatory bowel disease (including ulcerative colitis and Crohn's Disease), systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis), CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis). Patients with Graves disease and vitiligo will be allowed.
20. Patients with a history of a malignancy other than the one evaluated in this study enrollment, with exception of the following circumstances:

    * Patients with a history of malignancy who have been adequately treated and have been disease-free for at least 1 year, and
    * Patients with adequately treated active non-invasive cancers (such as non-melanomatous skin cancer or in-situ bladder, cervical and breast cancers).
21. Patients with psychiatric/social situations or addictive disorders that may compromise the ability of the patients to give informed consent or to comply with the study procedures.
22. Female patients who are pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of Dose-limiting toxicities (DLT) during the study treatment until 3 weeks after first NKR-2 study treatment administration. | during the study treatment until 3 weeks after first NKR-2 study treatment administration.
  Dose-limiting toxicity refers to a specific adverse event that is experienced during treatment and until 3 weeks after first NKR-2 dose administration, is new and at least possibly related to NKR-2 study treatment administered following a preconditioning regimen

SECONDARY OUTCOMES:
The NKR-2 cell kinetics endpoint of this Phase I study is: The evaluation of the circulating NKR-2 peripheral blood kinetics post-administration. | From day 1 (visit 4) until the end of the administration phase (day 85 = week 12 = Visit 22).
  NKR-2 detection in peripheral blood-isolated PBMC will be mandatory performed until the end of the administration phase. If positive at this visit, the evaluation will be performed during the follow-period visits and until 2 sequential tests are providing "undetectable" results, suggesting a lack of the NKR-2 persistence.
Additional Safety Endpoint: the occurence of Adverse Events ans Serious Adverse Events and any toxicity linked to study participation until the end of the administration phase, and until the end of the treatment follow-up | Until the end of the administration phase, and until the end of the treatment follow-up (at Month 24 - Visit 34).
  The occurrence of AEs and SAEs and any toxicity linked to study participation until the end of the administration phase, and until the end of the treatment follow-up (at Month 24 - Visit 34).
Clinical activity secondary endpoints: The incidence of CR, CRMRD-, CRi, MLFS, PR, or SD for AML patients. | From week 5 until Month 24.
  The incidence of CR, CRMRD-, CRi, MLFS, PR, or SD for AML patients at Week 5, Week 12, Week 19, Month 6, Month 9, Month 12, Month 18 and Month 24 post the first NKR-2 administration,
Clinical activity secondary endpoints: The incidence of CR, PR, marrow CR, cytogenic response, hematologic improvement or SD for MDS patients | From week 5 until Month 24.
  The incidence of CR, PR, marrow CR, cytogenic response, hematologic improvement or SD for MDS patients at Week 5, Week 12, Week 19, Month 6, Month 9, Month 12, Month 18 and Month 24 post the first NKR-2 administration
Clinical activity secondary endpoints: The objective clinical response rate (ORR) post the first NKR-2 administration | From week 5 until Month 24.
  The objective clinical response rate (ORR) post the first NKR-2 administration
Clinical activity secondary endpoints:The duration of response for patients with objective clinical response | From week 5 until Month 24.
  The duration of response for patients with objective clinical response
Clinical activity secondary endpoints: The ORR among subjects retreated with NKR-2. | From week 5 until Month 24.
  The ORR and duration of second response among subjects retreated with NKR-2.
Clinical activity secondary endpoints: The duration of second response among subjects retreated with NKR-2. | From week 5 until Month 24.
  The ORR and duration of second response among subjects retreated with NKR-2.
Clinical activity secondary endpoints: The overall survival (OS) from the study enrollment. | From study enrollment until Month 24.
  The overall survival (OS) from the study enrollment.
Clinical activity secondary endpoints: The relapse-free survival (RFS) from the study enrollment | From study enrollment until Month 24.
  The relapse-free survival (RFS) from the study enrollment
Clinical activity secondary endpoints: The event-free survival (EFS) from the study enrollment. | From study enrollment until Month 24.
  The event-free survival (EFS) from the study enrollment.
Clinical activity secondary endpoints: The cumulative incidence of relapse (CIR) | From study enrollment until Month 24.
  The cumulative incidence of relapse (CIR)
Clinical activity secondary endpoints: The cumulative incidence of death (CID) | From study enrollment until Month 24.
  The cumulative incidence of death (CID)
Clinical activity secondary endpoints: The non-relapse mortality (NMR) rate. | From study enrollment until Month 24.
  The non-relapse mortality (NMR) rate.
Mandatory correlative studies of this study are: The NKR-2 kinetics post-injection in the bone marrow. | From week 5 until month 24
  The aim of this specific research is to identify the presence of NKR-2 within and its kinetics post-administration according to the dose and preconditioning chemotherapy regimen. Genomic DNA isolated from these samples will be evaluated by qPCR using a validated assay (VCN) that detects a DNA signature unique to the NKR-2 transgene.
Mandatory correlative studies of this study are: Characterization of systemic cytokine level release post NKR-2 administration. | From day 1 until day 134 (week 19)
  One of the key effector functions of NKR-2 is the release of soluble cytokines during antigen engagement. Consequently, a surrogate marker of NKR-2 in vivo activity is potentially raised levels of cytokines relevant to T cell activation within the peripheral circulation.
Mandatory correlative studies of this study are: The evaluation of NKG2D ligand expression in patients' tumor cells prior to and after treatment. | From day 1 until day 134 (week 19)
  The research will evaluate NKG2D ligand expression in patient tumor samples. The aim of this project is to establish whether a correlation can be drawn between with the level of NKG2D ligand tumoral expression and NKR-2 activity.
Mandatory correlative studies of this study are: The evaluation of NKG2D ligand expression in patients' peripheral mononuclear cells prior to and after treatment. | From day 1 until day 134 (week 19)
  The research will evaluate NKG2D ligand expression in patient normal cells pre/post preconditioning chemotherapy and NKR-2 administrations. The aim of this project is to establish whether chemotherapy induce expression of NKG2D ligand expression and the possible correlation to any potential toxicity of the NKR-2 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Lehmann, MD, Study Director — Celyad Oncology SA
Locations (7):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Inc.,, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - New York School of Medicine, New York, New York
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Institute Jules Bordet, Brussels
  - UZ Gent, Ghent

IPD SHARING:
Plan to Share IPD: No